CLINICAL TRIAL: NCT03055039
Title: Epidemiology of New Born Child Pain in the Delivery Room
Brief Title: Epidemiology of Pain in the Delivery Room
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EPIDROOM
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: New Born Child Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The nociceptif system of the newborn child is functional from 22 to 23 weeks of pregnancy. During the delivery the baby is exposed to multiple exterior factors and he is capable to memorize the pain .Recent epidemiologic studies showed that the coverage of pain was insuffcient and also an increase of analgesic means. Normally the pain coverage have to be managed and group every painful gesture. In fact all these recommandations are not followed by medical team.

The aim of the study is to evaluate the prevalence of this type of pain as to set up an adequate coverage.

ELIGIBILITY:
Inclusion Criteria:

* Newborn child been born after 24 weeks amenorrheas undergoing a painful gesture in delivery room

Exclusion Criteria:

* Newborn child been born in palliative care
* non francophone parents

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn child been born after 24 weeks amenorrheas undergoing a painful gesture in delivery room
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of prevalence of the newborn child 's pain in delivery room | Day 1
  Counting the number of painful gesture (injection,blood test...)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No